CLINICAL TRIAL: NCT04509453
Title: Comparison Between McGRATH and Macintosh Laryngoscopy in Laryngeal Mask Airway Insertion
Brief Title: McGRATH vs Macintosh Laryngoscopy Comparison in LMA Insertion
Acronym: GRAN-PALM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Christopher Ryalino, Principal Investigator, Udayana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UNUD-CTR-FK270720-003; 1320/UN14.2.2.VII.14/LT/2020 (Other: Committee of Ethical Research of Udayana University)
Record Dates: First submitted 2020-07-27; First posted 2020-08-12 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Intubation Complication; Intubation;Difficult; Anesthesia
Keywords: successful intubation; classic LMA; video laryngoscopy; difficulty; cuff pressure leak

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- McGRATH (Experimental)
  Interventions: Device: McGRATH laryngoscopy; Device: Macintosh laryngoscopy
- Macintosh (Active Comparator)
  Interventions: Device: McGRATH laryngoscopy; Device: Macintosh laryngoscopy

INTERVENTIONS:
Device: McGRATH laryngoscopy — Patients who underwent general anesthesia with LMA insertion by using McGRATH video layngoscopy
  Other Names: Group G
Device: Macintosh laryngoscopy — Patients who underwent general anesthesia with LMA insertion by using classic Macintosh video layngoscopy
  Other Names: Group I

SUMMARY:
Various techniques have been developed to get a good LMA position, one of them is using a laryngoscope. The most popular laryngoscope used for LMA installation is the Macintosh type. Technological developments have brought laryngoscopes into the video era, one of which is McGRATH's laryngoscope, which from several studies about having an advantage in terms of the first attempt, time, complications, and hemodynamic stability of intubation. It needs to be proven through research on the comparison of clinical outcomes of LMA installation with McGrath laryngoscope and Macintosh laryngoscope.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent surgery with general anesthesia by LMA insertion in Sanglah General Hospital
* Agreed to be included in the study by signing informed consent
* American Society of Anesthesiologist physical status 1-2

Exclusion Criteria:

* Patients unfit for LMA insertion
* Patients with suspected airway management difficulty
* Pregnancy
* Morbid obese

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with first-attempt success | immediately after LMA insertion
  Successful LMA insertion within first attempt
Mean arterial pressure | immediately after LMA insertion
  Mean arterial pressure measured by non-invasive blood pressure monitor
Heart rate | immediately after LMA insertion
  Heart rate measured by standard monitor

SECONDARY OUTCOMES:
Time required | immediately after LMA insertion
  Time required for LMA insertion using the respective method
Complications | An hour after the the end of surgery
  Incidence of hoarseness or throat pain due to LMA insertion

CONTACTS AND LOCATIONS:
Locations (1):
- Sanglah General Hospital, Denpasar, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: No